CLINICAL TRIAL: NCT01724918
Title: Lacosamide IV and EEG/EKG (LIVE) Study
Acronym: LIVE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Time limitation for recruitment exceeded. 72 of 90 estimated sample recruited.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: UCB Pharma GmbH (Industry)
Responsible Party: Principal Investigator, Rick McLachlan, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LIVE 001
Record Dates: First submitted 2012-10-31; First posted 2012-11-12 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Focal Epilepsy
Keywords: IV lacosamide; focal epilepsy; EEG; EKG
MeSH Terms: conditions — Epilepsies, Partial | interventions — Lacosamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 100 mg IV (Other): 100 mg IV lacosamide infused over 30 minutes
  Interventions: Drug: Lacosamide
- 200 mg IV (Other): 200 mg IV lacosamide infused over 30 minutes
  Interventions: Drug: Lacosamide
- 400 mg IV (Other): 400 mg IV lacosamide infused over 30 minutes
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide
  Other Names: Vimpat

SUMMARY:
The purpose of this study is to evaluate the effect of different intravenous doses (IV) of a new anti-epileptic drug (AED) called lacosamide on continuous EEG (electroencephalogram) rhythms (or brain rhythms) in subjects with focal seizures and the tolerability of those doses by patients. In addition, this study will assess the effect of IV lacosamide on EKG (electrocardiogram), a test which checks for problems with the electrical activity of the heart.

DETAILED DESCRIPTION:
The impact of antiepileptic drugs on the EEG can vary from marked to none. A small number of AEDs also affect the EKG. Lacosamide is a new AED that selectively enhances slow inactivation of voltage-gated sodium channels, resulting in stabilization of hyperexcitable neuronal membranes and inhibition of repetitive neuronal firing. Information is lacking about the effect of lacosamide on brain and heart rhythms.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is informed and given ample time and opportunity to think about her/his participation and has given her/his written informed consent.
2. Adult patients 18-65 years
3. Diagnosis of focal epilepsy
4. Continuous EEG and video monitoring
5. Continuous EKG
6. Active EEG showing frequent spikes, electrographic or clinical seizures

Exclusion Criteria:

1. Subject has no IV access.
2. Subject is hemodynamically unstable.
3. Previous use of Lacosamide
4. Primary generalized epilepsy
5. Non-epileptic seizures
6. No significant cardiac, renal or hepatic disease
7. No cardiac arrhythmias including heart block
8. Subject is a pregnant or lactating woman.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-05; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in the number of interictal spikes | One hour before and after drug

SECONDARY OUTCOMES:
Change in frequency and quantity of background EEG rhythms | One hour before and after drug
Change in EKG (QT, PR interval and heart rhythm) | One hour before and after drug

OTHER OUTCOMES:
Adverse events | Up to 4 hours after start of infusion

CONTACTS AND LOCATIONS:
Overall Officials: Richard McLachlan, MD, FRCPC, Principal Investigator — London Health Sciences Centre, University Campus
Locations (4):
- Canada (4):
  - Foothills Medical Center, Calgary, Alberta
  - London Health Sciences Centre, London, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Royal University Hospital, Saskatoon, Saskatchewan